CLINICAL TRIAL: NCT03107754
Title: Buffered Lidocaine for Paracervical Block to Decrease Injection Pain During First Trimester Uterine Aspirations
Brief Title: Buffered Lidocaine in Paracervical Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-00083
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Results first posted 2020-05-15 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine; Anesthesia, Obstetrical

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A statistician not involved with the conduct of the study will use a computer random number generator to generate random permuted blocks. This statistician will place allocation assignment cards in sequentially numbered, sealed, opaque envelopes. A different randomization scheme will be used for each location, one at the Kapi'olani office and one at the Queen's office.
  A clinic staff member not involved with the conduct of the study will be trained specifically in the opening of the allocation envelopes. The staff member will be trained to open the envelope and remove the study card to read the allocation group: buffered lidocaine or plain lidocaine. The clinic staff member will then prepare the buffered lidocaine or plain lidocaine in an unlabeled syringe, and place it on the surgical tray.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard paracervical block (Placebo Comparator): A paracervical block will be administered with 20 cc of 1% lidocaine, which is our standard office protocol
  Interventions: Drug: Lidocaine
- Buffered lidocaine paracervical block (Experimental): A paracervical block will be administered with 20 cc of 1% lidocaine buffered with 8.4% sodium bicarbonate
  Interventions: Drug: Lidocaine-Sodium Bicarbonate

INTERVENTIONS:
Drug: Lidocaine — Paracervical block will be injected at 2 points at the cervicovaginal junction to decrease pain
  Other Names: Paracervical anesthesia
  Arms: Standard paracervical block
Drug: Lidocaine-Sodium Bicarbonate — Paracervical block will be injected at 2 points at the cervicovaginal junction to decrease pain
  Other Names: Buffered paracervical anesthesia
  Arms: Buffered lidocaine paracervical block

SUMMARY:
For pain relief during a first trimester surgical aspiration, most providers use the paracervical block, either alone or in combination with other pain control techniques. Some providers use buffered lidocaine due to a belief that it decreases pain. Others use plain lidocaine. At our clinics, the standard pain management protocol is using 20 cc of 1% plain lidocaine in a two site injection. Few studies have compared buffered versus unbuffered lidocaine for paracervical blocks during first trimester uterine aspirations. This study seeks to determine if buffered lidocaine decreases injection pain versus plain lidocaine for paracervical blocks.

DETAILED DESCRIPTION:
Potential participants will be identified at their office visits to the University Women's Health Specialists. If a patient desires uterine aspiration of a first trimester pregnancy or management of a failed pregnancy in the first trimester, they will first receive standard counseling. Only after providing written informed consent for the procedure will the patient's be screened for eligibility for our study. If the patient is eligible, she will be asked by a member of the research team if she is interested in participating. If she is, the study will be explained to her and written consent will be obtained after she is given the opportunity to have all of her questions answered. The patient will then complete a written questionnaire to collect demographic data.

This prospective randomized control trial will consist of two study arms. Participants will be randomly assigned to Arm 1, where a paracervical block will be administered with 20 cc of 1% lidocaine, which is our standard office protocol, or to Arm 2, where a paracervical block will be administered with 20 cc of 1% lidocaine buffered with 8.4% sodium bicarbonate. Prior to the start of the study, study assignments will be generated in a 1:1 ratio.

All patients who consent to the study will receive standard counseling prior to their procedure. The procedure will start with a bimanual exam by the provider. Next, the provider will place a speculum, cleanse the cervix with betadine solution, and place a single-tooth tenaculum on the anterior lip of the cervix. At this point, participants assigned to Arm 1 will receive a paracervical block loaded with 20 cc of 1% lidocaine and injected at 2, 4, 8 and 10 o'clock positions of the cervicovaginal junction. Participants assigned to Arm 2 will receive a paracervical block loaded with 18 cc of 1% lidocaine and 2 cc of 8.4% sodium bicarbonate and inject the block in the same fashion. The research assistant will ask the patient to verbally report their level of pain based on the 100 mm visual analog scale (VAS) at the following points of the procedure:

1. Prior to the start of the procedure (baseline anxiety)
2. After speculum placement
3. After paracervical block
4. After cervical dilation
5. After suction curettage
6. At end of procedure

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 14 years and older
* Desiring uterine aspiration for pregnancy or surgical management of a miscarriage
* Gestational age up to 13 weeks and 6 days to be established by best dating (i.e. last menstrual period or earliest ultrasound)
* Treatment plan involves outpatient uterine aspiration
* Participant able to provide informed consent in English and willing to participate in the study

Exclusion Criteria:

* Unable to read, speak, or understand English
* Unable to provide informed consent
* Currently incarcerated
* Under the age of 14 years
* Contraindications to receiving lidocaine or buffered lidocaine

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — University of Hawaii
Locations (1):
- Womens Options Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wiebe ER, Rawling M. Pain control in abortion. Int J Gynaecol Obstet. 1995 Jul;50(1):41-6. doi: 10.1016/0020-7292(95)02416-a. PMID 7556858
- [Background] Renner RM, Jensen JT, Nichols MD, Edelman AB. Pain control in first-trimester surgical abortion: a systematic review of randomized controlled trials. Contraception. 2010 May;81(5):372-88. doi: 10.1016/j.contraception.2009.12.008. Epub 2010 Jan 27. PMID 20399943
- [Background] Renner RM, Nichols MD, Jensen JT, Li H, Edelman AB. Paracervical block for pain control in first-trimester surgical abortion: a randomized controlled trial. Obstet Gynecol. 2012 May;119(5):1030-7. doi: 10.1097/AOG.0b013e318250b13e. PMID 22525915
- [Background] Renner RM, Edelman AB, Nichols MD, Jensen JT, Lim JY, Bednarek PH. Refining paracervical block techniques for pain control in first trimester surgical abortion: a randomized controlled noninferiority trial. Contraception. 2016 Nov;94(5):461-466. doi: 10.1016/j.contraception.2016.05.005. Epub 2016 May 25. PMID 27235677
- [Background] Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. Ann Emerg Med. 1996 Apr;27(4):485-9. doi: 10.1016/s0196-0644(96)70238-x. PMID 8604867
- [Background] Wiebe ER. Comparison of the efficacy of different local anesthetics and techniques of local anesthesia in therapeutic abortions. Am J Obstet Gynecol. 1992 Jul;167(1):131-4. doi: 10.1016/s0002-9378(11)91645-7. PMID 1442914
- [Background] Welch MN, Czyz CN, Kalwerisky K, Holck DE, Mihora LD. Double-blind, bilateral pain comparison with simultaneous injection of 2% lidocaine versus buffered 2% lidocaine for periocular anesthesia. Ophthalmology. 2012 Oct;119(10):2048-52. doi: 10.1016/j.ophtha.2012.05.029. Epub 2012 Jul 6. PMID 22771049
- [Background] Kizer NT, Zhao Q, Peipert JF, Ioffe Y, Massad LS. A randomized trial of buffered versus nonbuffered lidocaine with epinephrine for cervical loop excision. J Low Genit Tract Dis. 2014 Jan;18(1):8-12. doi: 10.1097/LGT.0b013e31828deffd. PMID 23774079
- [Background] Narvaez J, Wessels I, Bacon G, Chin VR, Baqai WK, Zimmerman GJ. Prospective randomized evaluation of short-term complications when using buffered or unbuffered lidocaine 1% with epinephrine for blepharoplasty surgery. Ophthalmic Plast Reconstr Surg. 2010 Jan-Feb;26(1):33-5. doi: 10.1097/IOP.0b013e3181b80c13. PMID 20090482
- [Background] Hobeich P, Simon S, Schneiderman E, He J. A prospective, randomized, double-blind comparison of the injection pain and anesthetic onset of 2% lidocaine with 1:100,000 epinephrine buffered with 5% and 10% sodium bicarbonate in maxillary infiltrations. J Endod. 2013 May;39(5):597-9. doi: 10.1016/j.joen.2013.01.008. Epub 2013 Mar 20. PMID 23611375
- [Background] Harreld TK, Fowler S, Drum M, Reader A, Nusstein J, Beck M. Efficacy of a Buffered 4% Lidocaine Formulation for Incision and Drainage: A Prospective, Randomized, Double-blind Study. J Endod. 2015 Oct;41(10):1583-8. doi: 10.1016/j.joen.2015.06.017. Epub 2015 Aug 4. PMID 26253800

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Paracervical Block | Buffered Lidocaine Paracervical Block
Started | 48 | 50
Completed | 48 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Paracervical Block: A paracervical block will be administered with 20 cc of 1% lidocaine, which is our standard office protocol
  Lidocaine: Paracervical block will be injected at 4 points at the cervicovaginal junction to decrease pain
- Buffered Lidocaine Paracervical Block: A paracervical block will be administered with 20 cc of 1% lidocaine buffered with 8.4% sodium bicarbonate
  Lidocaine-Sodium Bicarbonate: Paracervical block will be injected at 4 points at the cervicovaginal junction to decrease pain
- Total: Total of all reporting groups
Arm/Group | Standard Paracervical Block | Buffered Lidocaine Paracervical Block | Total
Number analyzed (Participants) | 48 | 50 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (6) | 28 (6) | 29 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 50 | 98
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants were allowed to select more than one ethnicity.
  Participants
    White/Caucasian | 18 | 17 | 35
    Black/African American | 3 | 2 | 5
    Asian | 26 | 31 | 57
    Native Hawaiian/Pacific Islander | 23 | 22 | 45
    American Indian/Alaska Native | 3 | 2 | 5
    Hispanic/Latino | 5 | 4 | 9
    Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Injection Pain
Description: For the primary outcome, pain immediately after paracervical block injection was measured by a scale. The scale used was the 100-mm visual analog scale. The minimum score was 0 and the maximum score was 100. Higher numbers indicate worse pain.
Time Frame: Immediately after injection of the paracervical block
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Paracervical Block | Buffered Lidocaine Paracervical Block
Number analyzed (Participants) | 48 | 50
units on a scale | 44.5 [18.25 to 65] | 30 [15.25 to 64.5]

2. Secondary Outcome: Pain After Speculum Placement, Cervical Dilation, and Aspiration
Description: Pain scores were measured at multiple points throughout the procedure. Pain scores were measured using a 100 mm visual analog scale with 0 being no pain and 100 being the worst pain ever.
Time Frame: Immediately after speculum placement, cervical dilation, uterine aspiration
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Standard Paracervical Block | Buffered Lidocaine Paracervical Block
Number analyzed (Participants) | 48 | 50
units on a scale
  After insertion of speculum | 13 (20.7) | 17 (21.85)
  After cervical dilation | 60.06 (26.30) | 55 (29.57)
  After uterine aspiration | 67.5 (26.44) | 69 (28.54)

ADVERSE EVENTS:
Time Frame: Each patient was assessed for adverse events during their procedure, during their recovery time, and upon discharge from the clinic for an average of one week.
Arm/Group | Standard Paracervical Block | Buffered Lidocaine Paracervical Block
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/50
Other Adverse Events (participants affected / at risk) | 0/48 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT03107754/Prot_SAP_001.pdf